CLINICAL TRIAL: NCT01339416
Title: Clinical Adverse Events In HIV-Infected Patients
Brief Title: HIV Cohort Study At Johns Hopkins University, University of North Carolina at Chapel Hill and Vanderbilt University
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: Johns Hopkins University (Other); University of North Carolina, Chapel Hill (Other); Vanderbilt University (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4001106
Record Dates: First submitted 2011-03-16; First posted 2011-04-20 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV infected cohort: HIV infected patients in the HIV cohorts at the three participating hospitals

SUMMARY:
Human Immunodeficiency Virus (HIV) infected patients in the HIV registries of Johns Hopkins University, University of North Carolina and Vanderbilt University will be followed in the routine clinical care to estimate the rates of prespecified clinical events in this population.

DETAILED DESCRIPTION:
All patients identified in the HIV registries will be included without any sampling

ELIGIBILITY:
Inclusion Criteria:

* HIV infection.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV infected patients seeking treatment at Johns Hopkins University, Vanderbilt University and University of North Carolina at Chapel Hill
Sampling Method: Non-Probability Sample
Enrollment: 8202 (Actual)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001106&StudyName=HIV%20Cohort%20Study%20At%20Johns%20Hopkins%20University%2C%20University%20of%20North%20Carolina%20at%20Chapel%20Hill%20and%20Vanderbilt%20University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and analyzed retrospectively from 3 clinical sites in the United States of America (Johns Hopkins University, University of North Carolina at Chapel Hill and Vanderbilt University).
Groups:
- All Participants: Participants who were diagnosed with Human immunodeficiency virus (HIV) infection and received HIV care during January 1, 2000 through December 31, 2010 (574 weeks) with follow-up extended up to 31st December 2011 (up to 626 weeks).
Period: Overall Study
Arm/Group | All Participants
Started | 8202
Completed | 8202
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 8202
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [32 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2348
  Male | 5854

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Malignancies
Description: Incidence rate of malignancies was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual from the date of HIV care initiation at that institution or January 1, 2000 if in care prior to this date. Malignancies included acquired immunodeficiency syndrome (AIDS)-defining malignancies and non-AIDS defining malignancies. AIDS-defining malignancies included invasive cervical cancer, non-Hodgkin's lymphoma and kaposis sarcoma; non-AIDS defining malignancies included but not limited to Hodgkin's disease, lung cancer, liver cancer, anal cancer, melanoma of the skin, leukemia, renal cancer, and prostate cancer. Overall data for non-AIDS defining malignancies and individual data for AIDS-defining malignancies was reported. Incidence rate was computed as the number of events per 100 person-years.
Time Frame: Up to Week 626
Population: Analysis population included all participants enrolled in the study. Here, n=participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Number (95% Confidence Interval); unit: malignancies per 100 person-years
Arm/Group | All Participants
Number analyzed (Participants) | 8202
malignancies per 100 person-years
  Non-Hodgkin's lymphoma (n= 8202) | 0.30 [0.24 to 0.36]
  Kaposis sarcoma (n= 8202) | 0.27 [0.22 to 0.34]
  Invasive cervical cancer (n= 2348) | 0.02 [0.002 to 0.07]
  Non-AIDS-defining (n= 8202) | 0.62 [0.54 to 0.72]

2. Primary Outcome: Incidence Rate of Acquired Immunodeficiency Syndrome (AIDS)-Defining Opportunistic Infections
Description: Incidence rate of AIDS-defining opportunistic infections was calculated as the number of events divided by person-time. Only the first diagnosis of each event per participant was included. Person-time was calculated as the sum of all time contributed by each individual from the date of HIV care initiation at that institution or January 1, 2000 if in care prior to this date. Opportunistic infections were those that occurred on immune-compromised participants. AIDS-defining infections included: esophageal candidiasis; pneumocystes jiroveci; non-tuberculous mycobacterium infection; AIDS dementia complex; disseminated cryptococcosis; cytomegalovirus (all sites); wasting syndrome; toxoplasmosis; cytomegalovirus retinitis; mycobacterium tuberculosis; Progressive (Prog.) multifocal leukoencephalopathy; histoplasmosis; cryptosporidiosis; recurrent pneumonia; herpes simplex infection; extra-pulmonary coccidioidomycosis; salmonella septicemia; isosporiasis.
Time Frame: Up to Week 626
Population: Analysis population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: infections per 100 person-years
Arm/Group | All Participants
Number analyzed (Participants) | 8202
infections per 100 person-years
  Candida esophagitis | 2.04 [1.88 to 2.20]
  Pneumocystes jiroveci | 1.72 [1.58 to 1.86]
  Mycobacterium infection | 0.77 [0.68 to 0.88]
  AIDS dementia complex | 0.66 [0.58 to 0.76]
  Disseminated cryptococcosis | 0.38 [0.31 to 0.45]
  Cytomegalovirus | 0.37 [0.31 to 0.44]
  Wasting syndrome | 0.28 [0.23 to 0.35]
  Toxoplasmosis | 0.25 [0.20 to 0.31]
  Cytomegalovirus retinitis | 0.22 [0.17 to 0.28]
  Mycobacterium tuberculosis | 0.20 [0.16 to 0.26]
  Prog. multifocal leukoencephalopathy | 0.16 [0.12 to 0.20]
  Histoplasmosis | 0.15 [0.11 to 0.19]
  Cryptosporidiosis | 0.13 [0.09 to 0.18]
  Recurrent pneumonia | 0.06 [0.04 to 0.10]
  Herpes simplex virus | 0.06 [0.03 to 0.09]
  Extrapulmonary coccidiodomycosis | 0.006 [0.00 to 0.02]
  Salmonella septicemia | 0 [0 to 0.01]
  Isosporiasis | 0 [0 to 0.01]

3. Primary Outcome: Incidence Rate of Myocardial Infarction
Description: Incidence rate of myocardial infarction (MI) was calculated as the number of events divided by person-time. Only first diagnosis of the event per participant was included. Person-time was calculated as the sum of all time contributed by each individual from the date of HIV care initiation at that institution or January 1, 2000 if in care prior to this date.
Time Frame: Up to Week 626
Population: Analysis population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: MI per 100 person-year
Arm/Group | All Participants
Number analyzed (Participants) | 8202
MI per 100 person-year | 0.27 [0.21 to 0.33]

4. Primary Outcome: Incidence Rate of Liver Failure
Description: Incidence rate of liver failure was calculated as the number of events divided by person-time. Only first diagnosis of the event per participant was included. Person-time was calculated as the sum of all time contributed by each individual from the date of HIV care initiation at that institution or January 1, 2000 if in care prior to this date.
Time Frame: Up to Week 626
Population: Analysis population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: liver failure per 100 person-years
Arm/Group | All Participants
Number analyzed (Participants) | 8202
liver failure per 100 person-years | 0.16 [0.12 to 0.21]

5. Primary Outcome: Incidence Rate of Viral Encephalitis
Description: Incidence rate of viral encephalitis was calculated as the number of events divided by person-time. Only first diagnosis of the event per participant was included. Person-time was calculated as the sum of all time contributed by each individual from the date of HIV care initiation at that institution or January 1, 2000 if in care prior to this date. Viral encephalitis was defined as inflammation of the brain due to virus.
Time Frame: Up to Week 626
Population: Analysis population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: viral encephalitis per 100 person-years
Arm/Group | All Participants
Number analyzed (Participants) | 8202
viral encephalitis per 100 person-years | 0.003 [0.00 to 0.02]

6. Secondary Outcome: Incidence Rate of Rhabdomyolysis
Description: Incidence rate of rhabdomyolysis was calculated as the number of events divided by person-time. Only first diagnosis of the event per participant was included. Person-time was calculated as the sum of all time contributed by each individual from the date of HIV care initiation at that institution or January 1, 2000 if in care prior to this date. Rhabdomyolysis was a condition of muscle fibers breakdown.
Time Frame: Up to Week 626
Population: Analysis population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: rhabdomylosis per 100 person-years
Arm/Group | All Participants
Number analyzed (Participants) | 8202
rhabdomylosis per 100 person-years | 0.10 [0.07 to 0.14]

7. Secondary Outcome: Incidence Rate of Death
Description: Incidence rate of death was calculated as the number of events divided by person-time. Person-time was calculated as the sum of all time contributed by each individual from the date of HIV care initiation at that institution or January 1, 2000 if in care prior to this date. All-cause mortality was used for the analyses.
Time Frame: Up to Week 626
Population: Analysis population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: death per 100 person-years
Arm/Group | All Participants
Number analyzed (Participants) | 8202
death per 100 person-years | 3.81 [3.60 to 4.02]

ADVERSE EVENTS:
Description: Due to the retrospective observational nature of study individual adverse events (AEs) were not planned to be collected and reported but only the pre-defined AEs which are represented as clinical endpoints reported in the outcome measure section.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Designation of primary and secondary endpoints was based on study team's inputs, as the endpoints were not prioritized in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes